CLINICAL TRIAL: NCT02460783
Title: Intermittent Calorie Restriction, Insulin Resistance, and Biomarkers of Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150123; 15-AG-0123
Record Dates: First submitted 2015-05-30; First posted 2015-06-02 (Estimated); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-11-15

CONDITIONS: Alzheimer's Disease; Obesity; Diabetes Mellitus
Keywords: Biomarkers; Diabetes; Obesity; Dementia of the Alzheimer Type; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Alzheimer Disease; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-2 CR (Experimental): Healthy living diet for 5 days/week; Calorie Restriction (480 Kcal in the form of a shake) for 2 days/week.
  Interventions: Other: Boost (R) 5-2 diet
- Healthy Living Diet (Active Comparator): Healthy living diet for 7 days/week
  Interventions: Other: Healthy Living Diet

INTERVENTIONS:
Other: Boost (R) 5-2 diet — Regular diet for 5 days/week; Calorie Restriction (480 Kcal in the form of a shake) for 2 days/week. Supplement providing 240 Kcal per shake. Participant takes 2 shakes per calorie restriction day.
  Other Names: 5-2 Intermittent Fasting (IF)
  Arms: 5-2 CR
Other: Healthy Living Diet — Counseling and educational material on diet portion, consistency
  Arms: Healthy Living Diet

SUMMARY:
Background:

- Insulin removes sugar from the blood to use for energy. Insulin resistance means that cells may not respond to insulin normally. It can lead to serious diseases. Researchers want to see how diet affects insulin resistance, weight, and brain chemicals related to Alzheimer s disease.

Objectives:

- To compare two forms of diet and their effects on insulin resistance and the brain.

Eligibility:

- Women ages 55 70 with insulin resistance.

Design:

* This study requires 6 clinic visits over 9 12 weeks. Participants must fast before visits.
* Visit 1, screening:
* Medical history, physical exam, and blood and urine tests.
* Participants will get a wrist device to wear for 4 days.
* Visit 2:
* Weight and waist measurement.
* Blood drawn.
* Questionnaires and thinking tests.
* Lumbar puncture. Skin will be numbed and a needle inserted between bones in the back will remove <TAB>fluid.
* Participants will drink a nutrition shake. Blood will be taken 12 times over 4 <TAB>hours through a thin tube in <TAB>the arm.
* Brain MRI. Participants will lie on a table that slides in and out of a cylinder in a strong magnetic field. <TAB>They will have a coil on their head and may do tasks.
* Participants will get advice about healthy eating and be randomly put in one of 2 groups. One group will get <TAB>nutrition shakes to drink.
* Visits 3 5:
* Weight and waist measurements, vital signs, blood draw, and questionnaires.
* Between visits, participants will get a call or email to check how they are doing.
* Visit 6: Repeat of visit 1.
* Participants will wear the wrist device for 4 more days, have a follow-up contact, then the study is finished.

DETAILED DESCRIPTION:
Being overweight or obese can cause insulin resistance (IR), which is defined as reduced responsiveness to insulin by the cells of various tissues or organs. IR at midlife increases the risk of developing Alzheimer s disease (AD). We recently discovered novel biomarkers of brain IR (altered Tyr and Ser phosphorylated forms of insulin receptor substrate 1; IRS-1) in plasma exosomes enriched for neuronal origin. Moreover, IR is associated with AD biomarkers including deficits in resting state brain activity and cognitive performance. Calorie restriction is defined as consuming fewer calories than what is considered normal without a lack of nutrients. A certain type of calorie restriction, in which one consumes 500-600 calories a day for two consecutive days, followed by non-restricted eating for 5 days (5-2 CR), has been shown to lower peripheral insulin resistance effectively. Effects of CR and lowering peripheral IR on brain IR and cognition are unknown. The goal of this exploratory pilot study is to provide proof-of-concept that 5-2 CR at midlife can reverse brain IR, lower peripheral IR, improve cognitive performance, and increase brain activation at rest and during tasks. Specifically, we will study the effects of 8 weeks of 5-2 CR versus a control dietary intervention on brain and peripheral IR, memory and executive function, resting state default mode network activity, brain metabolism, and AD biomarkers. Forty overweight to obese women and men (between 55 and 70 years of age) will be randomized 1:1 into 5-2 CR and control groups. In the 5-2 CR group, participants will be offered healthy living dietary counseling at baseline, which they will be instructed to implement for five days/week. For each of the other two consecutive days/week, they will consume two shakes (Boost , CWI Medical), providing a total of 480 Kcal/day. In the control group, participants will be offered healthy living dietary counseling at baseline, which they will be asked to implement for every day of the week. Participants will undergo screening including a history and physical examination, calculation of Body Mass Index (BMI, which must be greater than or equal to 27) and a blood draw for insulin and glucose to determine whether they have insulin resistance. If participants meet eligibility criteria, they will continue with a baseline visit involving anthropometric measures, questionnaires, tests of cognitive function, brain MRI, blood draws for plasma and peripheral blood mononuclear cells, and lumbar puncture for cerebrospinal fluid biomarkers of AD. After 8 weeks, we will collect the same measures. To assess and reinforce compliance with their respective diet, participants will come into the clinic every 2 weeks to discuss compliance, measure their body weight and perform blood draws for measurement of ketones to objectively confirm energy restriction for the 5-2 CR group. We will also contact participants every week to further ensure compliance. To assess the effects of the diets on physical activity, participants will be asked to wear an accelerometer for 96 hours before and after they are on the diet.

ELIGIBILITY:
* INCLUSION CRITERIA:
* BMI greater than or equal to 27; in addition, weight less than or equal to 350 lbs (weight limit for MRI scanner);
* Age of 55-70 years;
* HOMA-IR greater than or equal to 1.8;
* MMSE greater than or equal to 26

EXCLUSION CRITEIRA:

* History of clinically significant cardiovascular disease for the purpose of this study, such as chronic heart failure, coronary disease, cardiomyopathy, clinically significant cardiac valvular disease or clinically significant peripheral vascular disease. Cardiovascular conditions that are clinically non-significant for the purpose of this study, such as controlled hypertension, minor EKG abnormalities, mitral valve prolapse or benign murmurs are permissible;
* History of clinically significant stroke or other neurological disease of the central nervous system;
* History of substance abuse in the past 6 months or positive urine drug screen;
* History of clinically significant endocrine disorders (common mild endocrine disorders, such as untreated subclinical hypothyroidism with TSH < 10 mU/l or successfully treated hypothyroidism may be allowed);
* History of eating disorders, significant GI disorders or malabsorption disorders;
* History of type 2 diabetes; and/or use of anti-diabetes medications or insulin; and/or type 2 diabetes diagnosed during the screening visit based on fasting glucose > 125 mg/dL;
* History of hypoglycemia; and/or a fasting glucose < 70 mg/dL during the screening visit.
* Current use of systemic corticosteroids;
* Positive screening tests for HIV, HCV or HBV;
* Hematocrit less than 35% or hemoglobin less than 11 mg/dL;
* ALT or AST > 1.5 times the upper normal limit;
* Contraindications for MRI (pacemakers, ferrous metal implants or shrapnel in or around the head, etc.).
* Contraindications to LP, such as Coumadin, coagulopathy (international normalized ratio, or INR > 1.5; prothrombin time (PT), partial prothrombin time (PTT) > 1.5 x upper normal limit). Aspirin 81 mg qd is allowed. Aspirin up to 325 mg qd is allowed, if withheld for 7 days prior to the LP.
* Pregnancy or nursing.
* Refusal to consent to genetic testing for APOE.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios I Kapogiannis, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- [Derived] Kapogiannis D, Manolopoulos A, Mullins R, Avgerinos K, Delgado-Peraza F, Mustapic M, Nogueras-Ortiz C, Yao PJ, Pucha KA, Brooks J, Chen Q, Haas SS, Ge R, Hartnell LM, Cookson MR, Egan JM, Frangou S, Mattson MP. Brain responses to intermittent fasting and the healthy living diet in older adults. Cell Metab. 2024 Aug 6;36(8):1668-1678.e5. doi: 10.1016/j.cmet.2024.05.017. Epub 2024 Jun 19. PMID 38901423
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AG-0123.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 22 June 2015 and 23 December 2022.
Pre-assignment Details: 129 participants underwent screening; 80 were not eligible, 3 withdrew prior to randomization, and 46 participants were randomized, 22 to 5-2 CR and 24 to HL.
Period: Overall Study
Arm/Group | 5-2 CR | Healthy Living Diet
Started | 22 | 24
Completed | 20 | 20
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-2 CR | Healthy Living Diet | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (4.2) | 63.0 (6.1) | 63.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 7 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity was determined by self-report.
  Participants
    White/Caucasian | 14 | 11 | 25
    Black/African American | 6 | 8 | 14
    Hispanic | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 168.0 (9.2) | 168.0 (9.5) | 168.0 (9.2)
Body weight [Mean (Standard Deviation); unit: kg] | 99.0 (16.0) | 95.4 (10.7) | 97.2 (13.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.0 (4.0) | 33.8 (3.1) | 34.4 (3.6)
Homeostatic Model Assessment of Insulin Resistance 2 (HOMA2-IR) [Mean (Standard Deviation); unit: (μU/mmol/L)2] | 2.4 (0.7) | 2.3 (1.0) | 2.3 (0.9)
Mini-Mental State Examination (MMSE) score [Mean (Standard Deviation); unit: units on a scale] — Scores on the MMSE range from 0 to 30, with lower scores indicating greater impairment.
  units on a scale | 29.7 (0.6) | 29.3 (0.8) | 29.5 (0.7)
ApoE ε4 carrier status [Count of Participants; unit: Participants]
  Non-carrier | 17 | 12 | 29
  Carrier | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated Serine312-insulin Receptor Substrate-1 (pS312-IRS-1)
Description: IRS-1 is an intracellular adaptor molecule that is being recruited and activated by the binding of insulin and insulin-like growth factor to their respective receptors and in insulin resistance (IR) it shows aberrant phosphorylation in serine residues resulting in impaired downstream signal propagation. pS312-IRS-1 is considered an index of brain insulin resistance and a therapeutic response biomarker for interventions targeting brain IR. A decrease in its levels indicates target engagement with the intervention and improvement in brain IR.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | 79.01 (287.16) | 443.72 (182.56)
  Week 8 - Week 4 | -337.70 (256.08) | -608.92 (269.84)

2. Primary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) P-pan-Tyrosine-IRS-1 (pY-IRS-1)
Description: IRS-1 is an intracellular adaptor molecule that is being recruited and activated by the binding of insulin and insulin-like growth factor to their respective receptors and in insulin resistance (IR) it shows aberrant phosphorylation in tyrosine residues resulting in impaired downstream signal propagation. pY-IRS-1 is considered an index of brain insulin resistance and a therapeutic response biomarker for interventions targeting brain IR. A decrease in its levels indicates target engagement with the intervention and improvement in brain IR.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 5.05 (10.43) | 33.88 (32.28)
  Week 8 - Week 4 | -24.72 (10.76) | -54.23 (31.72)

3. Secondary Outcome: Mean Change in Body Weight
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
kg | -4.06 (0.72) | -2.33 (0.62)

4. Secondary Outcome: Mean Change in Body Mass Index (BMI)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
kg/m^2 | -1.41 (0.26) | -0.80 (0.20)

5. Secondary Outcome: Mean Change in Waist Circumference
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
cm | -2.84 (0.63) | -1.64 (0.82)

6. Secondary Outcome: Mean Change in Fasting Glucose
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | 0.57 (1.64) | 2.16 (1.64)

7. Secondary Outcome: Mean Change in Fasting Insulin
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: μIU/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
μIU/mL | -4.48 (1.08) | -2.87 (1.52)

8. Secondary Outcome: Mean Change in Homeostatic Model Assessment of Insulin Resistance 2 (HOMA2-IR)
Description: Homeostatic Model Assessment of Insulin Resistance Index 2 (HOMA2-IR) is a marker of peripheral insulin resistance and is calculated by fasting insulin (μIU/L) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance. A cut-off of 1.8 was used to indicate peripheral insulin resistance.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: μIU/L*mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
μIU/L*mg/dL | -0.49 (0.12) | -0.33 (0.18)

9. Secondary Outcome: Mean Change in Glycosylated Hemoglobin (HbA1c)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
percentage | -0.20 (0.08) | -0.02 (0.06)

10. Secondary Outcome: Mean Change in White Blood Cells (WBCs)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: cells x 10^9/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
cells x 10^9/L | -0.31 (0.23) | -0.23 (0.20)

11. Secondary Outcome: Mean Change in Red Blood Cells (RBCs)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: cells x 10^12/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
cells x 10^12/L | -0.12 (0.06) | -0.04 (0.05)

12. Secondary Outcome: Mean Change in Platelets
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: cells x 10^3/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
cells x 10^3/L | 2.18 (5.15) | 8.07 (4.10)

13. Secondary Outcome: Mean Change in Hemoglobin
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
g/dL | -0.29 (0.18) | -0.143 (0.15)

14. Secondary Outcome: Mean Change in Hematocrit
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
percentage | -1.08 (0.49) | -0.20 (0.39)

15. Secondary Outcome: Mean Change in International Normalized Ratio (INR)
Description: The International Normalized Ratio (INR) is derived from prothrombin time (PT) which is calculated as a ratio of the patient's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula: INR = Patient PT ÷ Control PT. The higher the INR, the longer it takes for blood to clot.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Ratio | 0.02 (0.01) | 0.02 (0.01)

16. Secondary Outcome: Mean Change in Serum Beta-Hydroxybutyrate (bHB)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mmol/L | 0.06 (0.03) | 0.03 (0.02)

17. Secondary Outcome: Mean Change in Serum Acetoacetate (AcAc)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mmol/L | 0.03 (0.01) | 0.01 (0.01)

18. Secondary Outcome: Mean Change in Serum Non-Esterified Fatty Acids (NEFA)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mEq/L | 0.09 (0.07) | 0.07 (0.04)

19. Secondary Outcome: Mean Change in Serum Cortisol
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
ng/mL | 22.89 (15.55) | 25.04 (12.63)

20. Secondary Outcome: Mean Change in Creatinine
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -0.01 (0.02) | -0.02 (0.02)

21. Secondary Outcome: Mean Change in Blood Urea Nitrogen (BUN)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -0.72 (1.04) | -0.55 (1.03)

22. Secondary Outcome: Mean Change in Alanine Aminotransferase (ALT)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
IU/L | -2.33 (1.45) | -0.77 (1.49)

23. Secondary Outcome: Mean Change in Aspartate Aminotransferase (AST)
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
IU/L | 0.87 (1.70) | 2.95 (2.49)

24. Secondary Outcome: Mean Change in Total Cholesterol
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -23.16 (6.17) | -16.29 (4.60)

25. Secondary Outcome: Mean Change in HDL Cholesterol
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -3.11 (1.34) | -4.01 (1.45)

26. Secondary Outcome: Mean Change in LDL Cholesterol
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -18.31 (5.82) | -11.59 (3.71)

27. Secondary Outcome: Mean Change in Triglycerides
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
mg/dL | -9.61 (6.72) | -6.61 (10.03)

28. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Amyloid Beta 42
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population). Measurements with coefficient of variation (CV) ≥ 20% were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | -43.56 (27.59) | -30.16 (36.70)

29. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Amyloid Beta 40
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | -608.42 (434.48) | -117.75 (565.04)

30. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Amyloid Beta 42 / Amyloid Beta 40 Ratio
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
Ratio | -0.0005 (0.001) | -0.004 (0.002)

31. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Total Tau
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | -13.45 (7.95) | -3.61 (4.12)

32. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) p181-Tau
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 13
pg/mL | -5.23 (10.67) | -1.82 (8.77)

33. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Neurogranin
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | 16.32 (9.25) | 2.70 (6.86)

34. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Light Chain Neurofilaments (Nf-L)
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | 134.31 (72.60) | 30.23 (26.86)

35. Secondary Outcome: Mean Change in Cerebrospinal Fluid (CSF) Glial Fibrillary Acidic Protein (GFAP)
Time Frame: Week 0, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 19 | 19
pg/mL | 1748.07 (1303.72) | 627.26 (624.30)

36. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Amyloid Beta 42
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -10.82 (25.178) | -9.58 (15.11)
  Week 8 - Week 4 | -0.62 (22.71) | 10.61 (17.28)

37. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Amyloid Beta 40
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -16.92 (23.41) | -4.84 (15.80)
  Week 8 - Week 4 | 11.47 (20.42) | 15.14 (20.20)

38. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Amyloid Beta 42 / Amyloid Beta 40 Ratio
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Ratio
  Week 4 - Week 0 | 0.01 (0.02) | -0.03 (0.02)
  Week 8 - Week 0 | -0.02 (0.02) | 0.01 (0.02)

39. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Total Tau
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -3.05 (25.93) | -5.33 (19.79)
  Week 8 - Week 4 | 8.00 (24.48) | 20.31 (26.43)

40. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) p181-Tau
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | 1.70 (15.72) | 1.01 (8.94)
  Week 8 - Week 4 | -1.65 (15.11) | 9.90 (12.26)

41. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) p231-Tau
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -3.47 (7.78) | -5.60 (4.71)
  Week 8 - Week 4 | -2.12 (7.10) | 0.13 (5.09)

42. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Akt
Description: Akt (or protein kinase B) is an insulin signaling cascade mediator. An increase in its levels indicates an improvement in brain insulin resistance.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 1.30 (2.79) | -3.27 (2.38)
  Week 8 - Week 4 | -2.15 (2.04) | -0.48 (2.93)

43. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated Serine473-Akt (pS473-Akt)
Description: pS473-Akt is an insulin signaling cascade mediator. An increase in its levels indicates activation of downstream insulin signaling pathway.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | -1.73 (1.80) | -5.13 (3.78)
  Week 8 - Week 4 | -3.33 (3.02) | -0.93 (4.00)

44. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated Serine473-Akt (pS473-Akt) / Akt Ratio
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Ratio
  Week 4 - Week 0 | -0.02 (0.02) | -0.01 (0.02)
  Week 8 - Week 4 | -0.01 (0.02) | -0.003 (0.02)

45. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated Extracellular Signal-regulated Kinase 1/2 (pERK1/2)
Description: pERK1/2 is an insulin signaling cascade mediator. An increase in its levels indicates activation of downstream insulin signaling pathway.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 4.66 (3.05) | -2.23 (2.82)
  Week 8 - Week 4 | -2.66 (2.90) | 0.37 (3.52)

46. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated c-Jun N-terminal Kinase (pJNK)
Description: JNK is an insulin signaling cascade mediator. Activated JNK (pJNK) inhibits insulin signaling. An increase in pJNK levels indicates inhibition of downstream insulin signaling pathway.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 2.91 (2.72) | -2.88 (3.30)
  Week 8 - Week 4 | -1.44 (3.08) | 8.44 (7.93)

47. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Phosphorylated p38 (pp38)
Description: p38 is an insulin signaling cascade mediator. Activated p38 (pp38) inhibits insulin signaling. An increase in pp38 levels indicates inhibition of downstream insulin signaling pathway.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 5.76 (7.10) | -1.39 (9.26)
  Week 8 - Week 4 | -12.20 (7.64) | 21.81 (25.47)

48. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) proBDNF
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -723.76 (814.01) | -91.37 (593.83)
  Week 8 - Week 4 | 531.01 (646.66) | -388.59 (984.13)

49. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) BDNF
Time Frame: Week 0, Week 4, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0: number analyzed (Participants) | 19 | 20
  Week 4 - Week 0 | 0.01 (1.22) | 1.07 (2.37)
  Week 8 - Week 4: number analyzed (Participants) | 20 | 19
  Week 8 - Week 4 | 0.98 (1.51) | 0.65 (3.09)

50. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Neurogranin
Time Frame: Week 0, Week 4, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0: number analyzed (Participants) | 20 | 19
  Week 4 - Week 0 | 5.69 (12.14) | 1.08 (14.91)
  Week 8 - Week 4 | -5.43 (12.50) | 4.07 (16.84)

51. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Heavy Chain Neurofilaments (Nf-H)
Time Frame: Week 0, Week 4, Week 8
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0: number analyzed (Participants) | 19 | 18
  Week 4 - Week 0 | -25.12 (47.07) | 4.80 (39.04)
  Week 8 - Week 4: number analyzed (Participants) | 18 | 17
  Week 8 - Week 4 | -1.59 (45.27) | 54.71 (56.18)

52. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) A-synuclein
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -4.21 (18.18) | -27.97 (9.23)
  Week 8 - Week 4 | 1.57 (13.87) | 17.06 (14.77)

53. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) TAR DNA-binding Protein 43 (TDP-43)
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
pg/mL
  Week 4 - Week 0 | -443.207 (324.78) | 67.84 (185.71)
  Week 8 - Week 4 | 64.67 (265.15) | 89.56 (258.47)

54. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Monocarboxylate Transporter 1 (MCT1)
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
ng/mL
  Week 4 - Week 0 | 158.32 (153.93) | -104.39 (167.54)
  Week 8 - Week 4 | -5.01 (139.56) | -141.72 (159.49)

55. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Monocarboxylate Transporter 2 (MCT2)
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
ng/mL
  Week 4 - Week 0 | 1.27 (1.14) | -1.72 (0.72)
  Week 8 - Week 4 | -0.67 (0.78) | 1.86 (1.37)

56. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Mitochondrial Complex IV Quantity
Description: Complex IV is part of the mitochondrial electron transport chain. Decreased complex IV levels in NDEVs have been found in patients with Alzheimer's disease. A decrease in its levels may indicate decreased ability of neurons for ATP production and energy crisis.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 0.00037 (0.00076) | -0.00006 (0.00035)
  Week 8 - Week 4 | -0.00051 (0.00047) | -0.00002 (0.00051)

57. Secondary Outcome: Mean Change in Neuron-Derived Extracellular Vesicle (NDEV) Mitochondrial Complex V Quantity
Description: Complex V is part of the mitochondrial electron transport chain. Decreased complex V levels in NDEVs have been found in patients with Alzheimer's disease. A decrease in its levels may indicate decreased ability of neurons for ATP production and energy crisis.
Time Frame: Week 0, Week 4, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units (AU)
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
Arbitrary Units (AU)
  Week 4 - Week 0 | 0.000082 (0.0002) | 0.00019 (0.0001)
  Week 8 - Week 4 | 0.00006 (0.00013) | -0.000074 (0.00036)

58. Secondary Outcome: Mean Change in Glucose by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Glucose concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Glucose relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population). Metabolite measurements with Cramer-Rao lower bounds (CRLBs) ≥ 20% were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.086 (0.034) | -0.013 (0.023)

59. Secondary Outcome: Mean Change in N-acetyl-aspartate by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) N-acetyl-aspartate concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. N-acetyl-aspartate relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.028 (0.034) | 0.054 (0.029)

60. Secondary Outcome: Mean Change in Lactate by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Lactate concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Lactate relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.016 (0.016) | -0.012 (0.012)

61. Secondary Outcome: Mean Change in Glutamate by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Glutamate concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Glutamate relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.014 (0.046) | 0.008 (0.047)

62. Secondary Outcome: Mean Change in Gamma-Aminobutyric Acid (GABA) by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Gamma-Aminobutyric Acid (GABA) concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Gamma-Aminobutyric Acid (GABA) relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 15
Ratio | 0.002 (0.023) | 0.020 (0.016)

63. Secondary Outcome: Mean Change in Glutamine by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Glutamine concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Glutamine relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.052 (0.029) | -0.004 (0.024)

64. Secondary Outcome: Mean Change in Glutathione by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Glutathione concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Glutathione relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.010 (0.010) | -0.018 (0.015)

65. Secondary Outcome: Mean Change in Myo-Inositol by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Myo-Inositol concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Myo-Inositol relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.046 (0.031) | -0.012 (0.028)

66. Secondary Outcome: Mean Change in N-acetyl-aspartyl-glutamate by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) N-acetyl-aspartyl-glutamate concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. N-acetyl-aspartyl-glutamate relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 11 | 17
Ratio | -0.038 (0.015) | 0.013 (0.016)

67. Secondary Outcome: Mean Change in Ascorbate by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Ascorbate concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Ascorbate relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 15 | 18
Ratio | -0.107 (0.050) | -0.076 (0.033)

68. Secondary Outcome: Mean Change in Alanine by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Alanine concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Alanine relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 17
Ratio | -0.006 (0.010) | -0.017 (0.010)

69. Secondary Outcome: Mean Change in Scyllo-Inositol by Proton J-PRESS MRS of Posteromedial Cortex (PMC)
Description: Proton J-PRESS Magnetic Resonance Spectroscopy (MRS) Scyllo-Inositol concentrations were determined using the Prior-Knowledge Fitting Procedure (ProFit), which fits linear combinations of simulated two-dimensional basis metabolite spectra. Scyllo-Inositol relative ratio to creatine was quantified.
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 11 | 13
Ratio | 0.002 (0.003) | 0.004 (0.004)

70. Secondary Outcome: Mean Change in Glucose by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 58
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | -0.002 (0.059) | 0.065 (0.040)

71. Secondary Outcome: Mean Change in Lactate by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 60
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 12 | 15
Ratio | 0.012 (0.019) | -0.017 (0.020)

72. Secondary Outcome: Mean Change in Glutamate by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 61
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | 0.010 (0.108) | -0.088 (0.056)

73. Secondary Outcome: Mean Change in Glutamine by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 63
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | -0.042 (0.046) | -0.048 (0.043)

74. Secondary Outcome: Mean Change in Glutathione by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 64
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | -0.011 (0.014) | 0.030 (0.018)

75. Secondary Outcome: Mean Change in Myo-Inositol by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 65
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | 0.001 (0.036) | -0.006 (0.035)

76. Secondary Outcome: Mean Change in N-acetyl-aspartyl-glutamate by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 66
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 12 | 12
Ratio | 0.001 (0.040) | 0.042 (0.026)

77. Secondary Outcome: Mean Change in Ascorbate by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 67
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 14 | 16
Ratio | -0.039 (0.075) | 0.006 (0.078)

78. Secondary Outcome: Mean Change in Alanine by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 68
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 13 | 16
Ratio | -0.009 (0.022) | 0.001 (0.021)

79. Secondary Outcome: Mean Change in Scyllo-Inositol by Proton J-PRESS MRS of Medial Prefrontal Cortex (MPFC)
Description: as for outcome 58
Time Frame: Week 0, Week 8
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 7 | 11
Ratio | -0.002 (0.008) | 0.004 (0.004)

80. Secondary Outcome: Mean Change in Executive Function Composite
Description: Executive function was assessed with the National Institutes of Health (NIH) Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER) battery that comprises written, verbal, and computerized tasks that test working memory, inhibition, set shifting, fluency, planning, insight, and social cognition and behavior. The Executive function Composite is a computerized score calculated based on the individual tests. It ranges between 0 and 10. Higher score values indicate better performance.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
units on a scale | 0.23 (0.05) | 0.07 (0.08)

81. Secondary Outcome: Mean Change in California Verbal Learning Test (CVLT)
Description: California Verbal Learning Test (CVLT) assesses verbal memory for unstructured information. Examinees are asked to recall words on a 16-item list after each of 5 learning trials (Immediate Free Recall; range 0-80 [5 x 0-16]). After a distractor list, participants are again asked to recall words spontaneously (Short Delay Free Recall; range 0-16) and with category cueing (Short Delay Cued Recall; range 0-16). Spontaneous recall (Long Delay Free Recall; range 0-16) and category cueing (Long Delay Cued Recall; range 0-16) are repeated after a 20-minute delay. Following the longer delay, participants also complete a yes/no recognition trial during which they need to discriminate between the target words and 32 distractor words (Long Delay Recognition; range 0-48 [0-16 true positive target words + 0-32 true negative distractor words]). Higher scores indicate better performance.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
units on a scale
  Immediate Free Recall | 4.55 (1.26) | 4.55 (1.13)
  Short Delay Free Recall | 0.75 (0.49) | 1.40 (0.65)
  Short Delay Cued Recall | 0.85 (0.33) | 0.75 (0.48)
  Long Delay Free Recall | 0.90 (0.48) | 0.10 (0.46)
  Long Delay Cued Recall | 1.40 (0.37) | 0.25 (0.44)
  Long Delay Recognition | 0.75 (0.58) | -0.35 (0.49)

82. Secondary Outcome: Mean Change in Logical Memory (LM) Test
Description: Logical Memory (LM) test assesses verbal memory for structured information. It consists of two thematically independent narrative stories. Each story has 25 items, which the examinee has to recall with as much detail and precision as possible. Each item is scored the same regardless of importance level, and all correct items are summed giving a maximum score of 25 for each story. "Verbatim recall" score only includes the items that are recalled exactly and with detailed information, whereas "gist recall" score includes both the verbatim recall and the items that are recalled with only the essential elements of the information. The examinee has to recall the two stories twice, immediately after their initial administration (immediate recall) and after a 20 to 30-minute delay (delayed recall). Total maximum score for each of the subtests is 50 (25 items x 2 stories) and the minimum score is 0. Higher scores indicate better performance.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
units on a scale
  Immediate Verbatim Recall | 1.60 (0.78) | 1.10 (0.95)
  Immediate Gist Recall | 1.65 (0.85) | 1.75 (1.04)
  Delayed Verbatim Recall | 1.30 (0.92) | 2.80 (1.26)
  Delayed Gist Recall | 1.95 (0.74) | 3.00 (1.35)

83. Secondary Outcome: Change in the Positive and Negative Affect Schedule (PANAS)
Description: Positive and Negative Affect Schedule (PANAS) is a 20-item self-report measure to assess positive and negative affect and is an index of emotional state. For positive affect, score can range from 10 - 50, with higher scores representing higher levels of positive affect. For negative affect, score can range from 10 - 50, with lower scores representing lower levels of negative affect.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
units on a scale
  Positive Affect | -2.45 (1.34) | -1.35 (0.96)
  Negative Affect | 0.51 (0.65) | -0.06 (0.57)

84. Secondary Outcome: Mean Change in the Short Form 36-item Health Survey (SF-36)
Description: Short Form 36-item Health Survey (SF-36) is a gauge of physical and psychosocial effects of the interventions. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability; the higher the score the less disability.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
units on a scale
  Physical functioning | 2.50 (2.49) | 2.00 (1.52)
  Role limitations due to physical health | 1.25 (3.74) | 0.00 (5.59)
  Role limitations due to emotional problems | -5.00 (3.56) | 0.00 (2.36)
  Energy/fatigue | 4.50 (3.35) | 3.75 (2.29)
  Emotional well-being | 1.00 (1.09) | 3.20 (1.73)
  Social functioning | 1.88 (2.21) | 0.00 (3.54)
  Pain | 3.00 (3.96) | 3.38 (3.19)
  General health | -2.25 (1.56) | -2.50 (1.79)

85. Secondary Outcome: Mean Change in Total Energy Expenditure
Description: Physical activity was monitored with an Actigraph GT3X-BT accelerometer device which measures accelerations in vertical, horizontal, and anterior-posterior directions.
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: kilocalories
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 19
kilocalories | -538.44 (626.72) | -302.86 (649.62)

86. Secondary Outcome: Mean Change in Daily Energy Expenditure
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: kilocalories/day
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
kilocalories/day | -18.76 (106.75) | -175.79 (113.50)

87. Secondary Outcome: Mean Change in Hourly Energy Expenditure
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: kilocalories/hour
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
kilocalories/hour | 0.23 (5.64) | -9.17 (5.86)

88. Secondary Outcome: Mean Change in Metabolic Rate
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: Watts/sec
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 19
Watts/sec | 0.01 (0.04) | -0.07 (0.04)

89. Secondary Outcome: Mean Change in Time in Activity
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 19
percentage of time
  Sedentary time | -0.013 (0.023) | 0.033 (0.021)
  Time in light physical activity | 0.008 (0.014) | -0.019 (0.012)
  Time in moderate physical activity | 0.005 (0.009) | -0.015 (0.010)
  Time in moderate-to-vigorous physical activity | 0.005 (0.009) | -0.015 (0.010)

90. Secondary Outcome: Mean Change in Total Steps
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: steps
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 19
steps | -4821.93 (2993.63) | -2937.65 (2362.82)

91. Secondary Outcome: Mean Change in Steps Per Minute
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: steps/minute
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 20
steps/minute | -0.13 (0.52) | -1.20 (0.67)

92. Secondary Outcome: Mean Change in Total Sedentary Bouts
Description: as for outcome 85
Time Frame: Week 0, Week 8
Population: FAS (full analysis set) is all randomized participants who completed 8 weeks of diet (per protocol population).
Measure: Least Squares Mean (Standard Error); unit: sedentary bouts
Arm/Group | 5-2 CR | Healthy Living Diet
Number analyzed (Participants) | 20 | 19
sedentary bouts | -17.69 (6.44) | 13.41 (5.49)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 5-2 CR | Healthy Living Diet
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-2 CR (N=20) | Healthy Living Diet (N=20)
Headache (General disorders) | 3 | 2
Lightheadedness (General disorders) | 1 | 0
Muscle cramps (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Loose stools (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02460783/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT02460783/ICF_001.pdf